CLINICAL TRIAL: NCT05636215
Title: A Phase 1/2, Multicenter, Open-label Study of IBI354 in Subjects with Locally Advanced Unresectable or Metastatic Solid Tumors
Brief Title: A First-in-human Study of IBI354 in Subjects with Locally Advanced Unresectable or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI354A101
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Unresectable or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI354 (Experimental): Single arm
  Interventions: Biological: IBI354

INTERVENTIONS:
Biological: IBI354 — Recombinant Anti-HER2 monoclonal Antibody-Camptothecin derivative conjugate for injection

SUMMARY:
This is a Phase 1/2, open-label, multicenter study designed to evaluate the safety, tolerability, and DLTs to establish the maximum tolerated dose (MTD) or maximum administered dose (MAD), and the RP2D of sequential doses of IBI354 (study drug), and to explore and confirm the efficacy, safety and tolerability of IBI354 in subjects with locally advanced unresectable or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ≥ 18 years
2. Phase 1a : Has a pathologically documented advanced/unresectable or metastatic solid tumor with HER2 alterations (IHC 1+, IHC 2+, IHC 3+ and/or ISH+ and/or NGS confirmed mutant or amplification).

   Phase 1b/2: Selected solid tumors enrolled Subjects with advanced GC/BC/BTC/CRC/Gyn with her2 expression (IHC 1+, IHC 2+, IHC 3+ and/or ISH+).
3. Adequate bone marrow and organ function
4. Subjects, both male and female, who are either not of childbearing potential or who agree to use at least one highly effective method of contraception during the study (begin from screening or within 2 weeks prior to the first dose, whichever comes first, and continue until 6 months after the last dose of study drug); Subjects, both male and female, who are either not of childbearing potential or who agree to use a highly effective method of contraception during the study beginning within 2 weeks prior to the first dose and continuing until 6 months after the last dose of study drug
5. Subjects with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
6. Have LVEF ≥ 50% by echocardiography (ECHO) within 28 days before study drug administration.

Exclusion Criteria:

1. Received previous anti-tumor therapy within 4 weeks or 5 half-lives of the anti-tumor regimens before the first administration of study drug, whichever is shorter;
2. Plan to receive other antitumor therapy during the study excluding palliative radiotherapy for the purpose of symptom (like pain) relief that must also do not have impact on tumor assessment throughout the study;
3. Potent cytochrome P450 3A4 (CYP3A4) inhibitors within 2 weeks or 5 half-lives (whichever is longer) before first administration of the study drug.
4. Has adverse reactions resulting from previous antitumor therapies, which have not resolved to Grade 0 or 1 toxicity according to NCI-CTCAE v5.0 (except for alopecia, fatigue, pigmentation and other conditions with no safety risk according to investigators' opinion) or baseline prior to first administration of the study drug;
5. Known symptomatic central nervous system (CNS) metastases.
6. History of pneumonia requiring corticosteroids therapy, or history of clinically significant lung diseases or who are suspected to have these diseases by imaging at screening period;
7. Uncontrolled diseases including:

   * Uncontrolled infection requiring systematic antibiotics, antivirals or antifungals within 2 weeks prior to first administration of the study drug;
   * Known human immunodeficiency virus (HIV) infection, or HIV positive (HIV 1/2 Ab positive);
   * HBsAg positive and/or HBcAb positive with HBV DNA titer ≥ 104 copies/mL or ≥ 2000 IU/mL or higher than lower limit of detection or HCV Ab positive with HCV RNA>103 copies/mL;
   * Active infection with COVID-19;
   * Active tuberculosis infection, or still on anti-tuberculosis therapy or received anti-tuberculosis therapy within 1 year prior to first administration of the study drug;
   * Active syphilis infection or latent syphilis requiring treatment;
   * Symptomatic congestive heart failure Grade II-IV, symptomatic or uncontrolled arrhythmias, QTc interval > 480 ms or personal or family history of congenital long/short QT syndrome;
   * SBP ≥ 160mmHg or DBP ≥ 100mmHg;
8. History of any arterial thromboembolic event within 6 months prior to the first administration of study drug, including myocardial infarction, unstable angina pectoris, cerebrovascular stroke or transient ischemic attack, etc.;
9. Risk of intestinal obstruction or perforation (including but not limited to: acute diverticulitis, abdominal abscess, etc.) or a history of inflammatory bowel disease, Crohn's disease, ulcerative colitis, or chronic diarrhea;
10. Do not have adequate treatment washout period before study drug administration, defined as:

    * Major surgery; ≥ 4 weeks.
    * Radiation therapy；≥ 4 weeks (if palliative stereotactic radiation therapy, ≥ 2 weeks).
    * Autologous transplantation；≥ 3 months.
    * Hormonal therapy；≥ 2 weeks.
    * Chemotherapy (including antibody drug therapy or other antitumor therapy)； ≥ 3 weeks.
    * Immunotherapy； ≥ 4 weeks.
    * Cytochrome P450 (CYP) 3A4 strong inhibitor；≥ 3 elimination half-lives of the inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs), treatment-emergent AEs (TEAEs). | Up to 30 days after the last administration
  An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. A TEAE will be defined as any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment has been administered.
Number of dose-limiting toxicity (DLT) | 21 days during the first cycle in Phase Ia
  Incidence of dose-limiting toxicity (DLT) events.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR).
duration of response (DoR) | Up to 2 years
  DoR is defined as the time from the date of first documented tumor response (CR/PR) until PD/death.
progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of first dose of study drug to the date of the first documented progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the date of first dose of study drug until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (4):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Sunshine Coast University Private Hospital, Sunshine Coast, Queensland
  - Monash Health, Clayton, Victoria
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No